CLINICAL TRIAL: NCT05202704
Title: Investigating the Hypoalgesic Effects of Spinal Manipulative Therapy Using Hidden Pain Conditioning and Positive Expectation in Chronic Low Back Pain Patients: Protocol for a Randomized Controlled Trial
Brief Title: Investigating the Hypoalgesic Effects of Manipulative Therapy Using Pain Conditioning and Expectations in Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Sao Carlos (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Thais Chaves, Associate Professor, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 52925921.5.0000.5504
Record Dates: First submitted 2021-12-03; First posted 2022-01-21 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Chronic Low Back Pain
Keywords: Placebo Effect; Contextual Effect; Spinal Manipulative Therapy; Expectations; Chronic Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental: Hidden conditioning procedure + Positive Expectation (Experimental): Patients with chronic low back pain will receive verbal delivered positive instructions regarding manipulative therapy. Then, after the spinal manipulative therapy they will be submitted to a hidden conditioning procedure in which the pain threshold will be surreptitiously downgrade to conditioning pain decrease to manipulative therapy (G1).
  Interventions: Procedure: Procedure/Surgery: Experimental: Hidden conditioning + Positive Expectation; Procedure: Spinal Manipulative Therapy
- Active Comparator: Positive expectations (Active Comparator): Patients with chronic low back pain will receive verbal delivered positive instructions regarding spinal manipulative therapy (G2) before the administration of a spinal manipulative therapy approach.
  Interventions: Procedure: Procedure/Surgery: Active Comparator: Positive Expectation; Procedure: Spinal Manipulative Therapy
- Active Comparator: Neutral Expectations (Active Comparator): Patients with chronic low back pain will receive verbal delivered neutral instructions regarding spinal manipulative therapy (G3) before the administration of a spinal manipulative therapy approach.
  Interventions: Procedure: Procedure/Surgery: Active Comparator: Neutral Expectation; Procedure: Spinal Manipulative Therapy

INTERVENTIONS:
Procedure: Procedure/Surgery: Experimental: Hidden conditioning + Positive Expectation — Patients will be submitted to quantitative sensory testing to determine different thresholds of noxious heat pain stimulus (intense, moderate or weak). Afterward, participants will receive instructions with the aim to induce positive expectations about the treatment by means of a workshop. Immediately after the first session of manipulative therapy, participants will be submitted again to the QST but now the heat pain threshold of the hidden conditioning group will be surreptitiously downgraded (the intense noxious stimulus will be downgraded to the moderate stimulus - individually obtained during the QST) as a mean to conditioning patients to believe that spinal manipulative therapy promoted pain relief. Patients will be invited to report the pain intensity perceived just after the QST (second test - conditioning procedure). The objective of questioning the pain intensity after the conditioning test is a procedure check to ensure that the conditioning procedure worked.
  Arms: Experimental: Hidden conditioning procedure + Positive Expectation
Procedure: Procedure/Surgery: Active Comparator: Positive Expectation — Patients in this group will be submitted to a quantitative sensory testing to determine different thresholds of noxious heat pain stimulus (intense, moderate or weak). Afterward, participants will receive instructions with the aim to induce positive expectation about the treatment by means of a workshop. Immediately after the first session of spinal manipulative therapy, participants will be submitted again to the QST (without downgrading of the intense noxious heat stimulus). Patients will be invited to report the pain intensity perceived during the QST after the intervention. The objective of questioning the pain intensity in this group is a procedure check - to investigate whether the positive instructions will show any effect.
  Arms: Active Comparator: Positive expectations
Procedure: Procedure/Surgery: Active Comparator: Neutral Expectation — Patients in this group will be submitted to a quantitative sensory testing to determine different thresholds of noxious heat pain stimulus (intense, moderate or weak). Afterward, participants will receive instructions with the aim to induce neutral expectation about the treatment by means of a workshop. Immediately after the first session of spinal manipulative therapy, participants will be submitted again to the QST (without downgrading of the intense noxious heat stimulus). Patients will be invited to report the pain intensity perceived during the QST after the intervention. The objective of questioning the pain intensity in this group is a procedure check - to investigate/confirm the effect of neutral instructions.
  Arms: Active Comparator: Neutral Expectations
Procedure: Spinal Manipulative Therapy — All the groups recruited in the study will receive five sessions of Spinal Manipulative Therapy. The intervention will be performed with the patient in the supine position. The clinician-researcher will passively lean over the patient to the side to be manipulated and ask the patient to place their hands behind their head. The researcher will then passively rotate the patient on the side to be manipulated and perform a posterior and inferior thrust on the opposite anterosuperior spine. The patients will receive 4 maneuvers (twice towards right side and twice towards left side).

SUMMARY:
The objective of this study will be to identify whether a conditioning procedure by the surreptitious downgrade of a noxious stimulus intensity associated with induced positive expectations about treatment will result in greater hypoalgesic effects when compared to positive verbal suggestions (positive expectation induction) alone regarding the effects of spinal manipulative therapy intervention in patients with CLBP. This study will enroll 264 individuals with CLBP aged between 18 and 60 years. Spinal Manipulative Therapy in the lumbar spine will be administered to all participants during 5 sessions.

First assessment session - participants will be submitted to a quantitative sensory testing (QST) to determine the heat pain threshold (calibration test) to run the conditioning procedure. Afterward, participants will be allocated by a blinded researcher into the following subgroups: hidden conditioning + positive expectation (G1); positive expectation alone (G2) and a group submitted to neutral expectations (G3) about the treatment.

First treatment session - Firstly, participants will receive instructions with the aim to induce positive (or neutral) expectations by means of a workshop. Secondly, all the participants will be submitted again to the pre-conditioning test, using the more intense pain stimulus obtained in the calibration test, then patients will be assessed regarding pain intensity and finally submitted to the manipulative therapy. At the end of the first treatment session, the conditioning test will be repeated, but the heat pain threshold of the hidden conditioning group (G1) will be surreptitiously downgraded (from intense pain stimulus to moderate pain stimulus) as a means of conditioning patients to believe that manipulative therapy promoted pain relief. Pain intensity will be assessed again to confirm a decrease in pain intensity.

Outcomes will be assessed three times: immediately after the five therapy sessions, one month later, and three months later. The primary outcomes assessed will be pain intensity and global perceived effect of improvement. The secondary outcome will be low back pain disability.

DETAILED DESCRIPTION:
Background: The term "contextual effect" has been used to reinforce the view that the placebo effect should be understood as an effect related to the therapeutic context, and not restricted to the use of inert treatments. Thus, the placebo effect is inherent to any therapeutic context and also can be used to enhance the effects of treatment with active components. There is evidence of the effectiveness of manipulative therapy in the treatment of chronic low back pain (CLBP), however, for most physical therapy interventions, its effect is small. Thus, strategies to enhance the effects of this therapy, such as through the use of context factors, may contribute to better therapeutic outcomes. The literature describes conditioning or positive induced expectation models to favor the placebo effect. Although some previous studies have shown that expectation alone or associated with conditioning procedures may intensify the hypoalgesic effects of therapies, no previous work has verified the isolated or associated hypoalgesic effect of conditioning and induction of expectancy on treatment in patients with CLBP undergoing manipulative therapy. Thus, the objective of this study will be to identify whether a conditioning procedure through surreptitious downgrade of nociceptive stimulus intensity associated with positive induced expectation about treatment will result in greater hypoalgesic effects when compared to positive verbal suggestions (expectations) induced or expectation alone regarding the effects of the Spinal Manipulative Therapy intervention in patients with CLBP. Methods: it will be a randomized controlled trial with a blinded assessor. It will be investigated the effect of the use of a hidden conditioning procedure and the induction of positive expectations on pain intensity after the administration of a manipulative therapy approach. We will enroll 264 patients with nonspecific CLBP aged 18 to 60 years will participate in this study. The sample size calculation was based on a minimal difference between groups of 2 units on pain intensity and overall perception of improvement (primary outcomes). All patients will undergo 5 sessions of Manipulative Therapy in the lumbar spine, except the no-treatment group (G3). In the first session, patients will be subjected to the inclusion and exclusion criteria and the calibration test (quantitative sensory testing) to determine the intense, moderate and weak thermal pain threshold, using the Q-sense equipment, for the conditioning procedure.

In the second session (beginning of the treatment), firstly the patients will be randomized to one of the three groups by a blinded assessor: hidden conditioning + positive expectations (G1) group; positive expectations group (G2) and neutral expectation group (G3). Following, participants will receive specific instructions to induce expectation in G1 and G2, and for G3, neutral instructions.

In the first treatment session - patients will receive the pre-conditioning test (heat pain), then they will be submitted to the manipulative therapy and again undergo the heat-conditioning post-testing. However, G1 will receive hidden conditioning (surreptitiously downgrade of noxious stimulus intensity from intense to moderate pain) to reinforce the association between manipulative therapy and pain intensity reduction. Pain intensity will be assessed just after the conditioning procedures as a manipulation check of the downgrading of the noxious stimulus.

The main hypothesis of this study is that the group undergoing hidden conditioning associated with positive induced expectation will have a higher hypoalgesic effect than the other groups immediately post-treatment.

Outcomes will be assessed three times: immediately after the five therapy sessions, one month later, and three months later. The primary outcomes assessed will be pain intensity and global perceived effect of improvement. The secondary outcome will be low back pain disability.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria for patients were as follows:

1. Patients who report non-specific CLBP (in which the specific nociceptive source cannot be identified, confirmed by a medical assessment) for at least three months duration;
2. Age ranged from 18 years to 60 years
3. Baseline pain intensity score ≥3 on a Numeric Pain Rating Scale (NPRS) (because of the measurement error > 2 reported for the NPRS);
4. Score greater than 14% on the Oswestry Disability Index (ODI) (to surpass the smallest detectable change of the ODI total score
5. Patients able to speak and understand Portuguese well to fill out the questionnaires.

Patients will be excluded if they met any of the following criteria:

1. Previous poor experiences with SMT through the application of a brief screening questionnaire
2. Pregnancy
3. Specific low back pain disorders like radiculopathy or lumbar stenosis or chronic degenerative disorders, i.e., uncontrolled cardiovascular, metabolic, or systemic diseases, neurological or psychiatric diseases, and stroke sequelae
4. Undergoing other therapeutic interventions for chronic pain and low back pain (including surgeries) in the last 3 months
5. Presence of contraindications to SMT
6. Patients who reach the upper limit of 50ºC, which is the maximum temperature provided by the Q-sense equipment described in the Medoc, Israel website

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 264 (Estimated)
Dates: Start 2022-02-20 (Actual); Primary Completion 2023-12-10 (Estimated); Study Completion 2024-03-10 (Estimated)

PRIMARY OUTCOMES:
Numeric pain rating scale (NPRS) | 6 weeks after randomization
  The NPRS used in this trial will consist of numbers from 0 to 10, in which 0 represents "no pain" and 10 represents "worst pain imaginable". High scores mean worse pain intensity.
Global Perceived Effect (GPE) | 6 weeks after randomization
  The GPE of improvement used for this trial is an 11-point scale that ranges from - 5 ("vastly worse") through 0 ("no change") to + 5 ("completely recovered") and participants are asked: "Compared to when this episode first started, how would you describe your orofacial pain these days?". A higher score indicates higher perception of recovery from the condition.

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) | 6 weeks and 3 months after randomization
  The ODI consists of 10 items, each of which has six response options. The total score will be calculated by summing up all the points, ranging from 10 to 50. This sum will be transformed into a percentage (0 to 100). High scores mean worse disability.

OTHER OUTCOMES:
Stanford Expectation Treatment Scale (SETS) | Baseline
  The scale contains six questions and seven answer alternatives, ranging from strongly disagree, partially disagree, slightly disagree, neither agree nor disagree, slightly agree, partially agree, and entirely agree to strongly disagree, partially disagree, slightly agree, partially agree, and fully agree. The positive expectation domain must include the total of items 1, 3 and 5 (score ranging from 7-21), while the negative expectation domain must include the sum of questions 2, 4 and 6 (score ranging from 7-21).
Low Back Pain Improvement Expectation Scale | Baseline
  The Scale evaluates a patient's past estimate that his or her low back pain would get better (regardless of the treatment used)."What are the chances of receiving relief from low back pain?" the participant will be asked.The participant will be given an 11-point scale to answer on, with 0 representing "no possibility" and 10 representing "extremely probable".
Patient Health Questionnaire-9 (PHQ-9) | Baseline
  The PHQ-9 Brazilian version will be used to assess symptoms of depression. Patients will be asked to rate nine questions on a four-point scale over the two weeks before to the administration of the questionnaire in this self-report measure. Validity has been assessed against an independent structured mental health professional interview. The PHQ-9 Brazilian version showed suitable structural validity (Confirmatory Fit Index = 0.98)
General Anxiety Disorder-7 (GAD-7) | Baseline
  The GAD-7 is a widely used diagnostic self-report scale for anxiety disorder screening, diagnosis, and severity assessment. Patients will be asked to rate their anxiety-related difficulties on a four-point scale over the two weeks before to the administration of the questionnaire in this self-report measure. GAD-7 scores vary from zero to 21, with higher GAD-7 scores being linked to more severe generalized anxiety. The psychometric properties of the GAD-7 in Brazilian Portuguese showed a one-dimensional structure and good internal consistency (α = 0.88). GAD-7 Brazilian version showed suitable internal consistency (Cronbach's alpha = .916) and reliability coefficient (ρ= .909).
Tampa Scale for Kinesiophobia (TSK) | Baseline
  TSK is a self-report questionnaire that assesses the fear of movement through 17 items that address pain and symptom intensity. The scores for each item range from 1 to 4 points (1 point for "strongly disagree", 2 points for "partially disagree", 3 points for "agree" and 4 points for "strongly agree"). For the total score, it is necessary to invert the scores of questions 4, 8, 12 and 16. The final score can range from 17 to 68 points, higher scores represent stronger beliefs about fear of movement.
Pain Catastrophizing Scale (PCS) | Baseline
  PCS is a self-administered questionnaire that consists of 13 items for the assessment of catastrophizing thoughts. It is divided into three domains: helplessness, magnification, and rumination. Each item is scored on a 5-point ordinal scale. The B-PCS total score ranges from 0 to 52 points, higher values denote greater pain catastrophizing. Acceptable values for validity, internal consistency, and test-retest reliability are described for the Brazilian PCS.
Positive and Negative Affect Scales (PANAS) | Baseline
  PANAS will be used to assess the positive and negative affect constructs. The scale is made up of 40 items, each factor made up of 20 adjectives that represent the subjects' moods and emotions. Each adjective is rated by the patients on a five-point Likert scale. The Brazilian Portuguese demonstrated acceptable measurement properties. The scale showed suitable internal consistency (Cronbach's Alpha = 0.84) and structural validity.
Pain Self-Efficacy Questionnaire (PSEQ) | Baseline
  Study patients will be evaluated on self-efficacy related to chronic pain, which can be defined as an individual's confidence that he/she can successfully produce desirable results related to living with chronic pain. The PSEQ has ten items which are rated on a seven-point ordinal. It was cross cultural adapted and validated to Brazilian Portuguese. Previous research showed an effect on self-efficacy using a pain neuroscience education intervention based on metaphors compared to an intervention using cognitive- behavioral concepts. PSEQ Brazilian version showed suitable internal consistency (Cronbach's alpha = .90) and construct validity when compared to Roland Morris Questionnaire (r=-.58).

CONTACTS AND LOCATIONS:
Overall Officials: Thais Chaves, PhD, Study Chair — Federal University of São Carlos - UFSCar
Locations (1):
- Unidade Saúde Escola - USE, São Carlos, São Paulo, Brazil

REFERENCES:
- [Derived] Nogueira Carrer HC, Lima TC, George SZ, Reis FJJD, Dias DLC, Campanha BES, Chaves TC. Investigating the hypoalgesic effects of spinal manipulative therapy using hidden pain conditioning and positive expectation in patients with chronic low back pain: protocol for a randomised controlled trial. BMJ Open. 2023 Apr 12;13(4):e066199. doi: 10.1136/bmjopen-2022-066199. PMID 37045570